CLINICAL TRIAL: NCT05751226
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Different Titration Schedules of Subcutaneous Doses of BI 1820237 Alone or Together With Either Semaglutide or BI 456906 in Otherwise Healthy Male and Female Individuals With Obesity/Overweight (Multiple Dose, Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in People With Overweight or Obesity to Test How Well Different Doses of BI 1820237 Are Tolerated When Given Alone or in Combination With Either Semaglutide or BI 456906
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1458-0002; 2022-002733-34 (EudraCT Number)
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide; BI 456906

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- BI 1820237 treatment group (Experimental)
  Interventions: Drug: BI 1820237
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 1820237 + semaglutide treatment group (Experimental)
  Interventions: Drug: BI 1820237; Drug: semaglutide
- placebo + semaglutide group (Active Comparator)
  Interventions: Drug: semaglutide; Drug: Placebo
- BI 1820237 + BI 456906 treatment group (Experimental)
  Interventions: Drug: BI 1820237; Drug: BI 456906
- placebo + BI 456906 group (Active Comparator)
  Interventions: Drug: Placebo; Drug: BI 456906

INTERVENTIONS:
Drug: BI 1820237 — BI 1820237
  Arms: BI 1820237 + BI 456906 treatment group; BI 1820237 + semaglutide treatment group; BI 1820237 treatment group
Drug: semaglutide — semaglutide
  Arms: BI 1820237 + semaglutide treatment group; placebo + semaglutide group
Drug: Placebo — Placebo
  Arms: Placebo group; placebo + BI 456906 group; placebo + semaglutide group
Drug: BI 456906 — BI 456906
  Arms: BI 1820237 + BI 456906 treatment group; placebo + BI 456906 group

SUMMARY:
This study is open to adults between 18 and 55 years of age who are living with overweight or obesity. People with a body mass index (BMI) from 27 to 40 kg/m2 can join the study.

The main purpose of this study is to find out how a medicine called BI 1820237 is tolerated by people with overweight or obesity when taken alone or in combination with a medicine called semaglutide or with a medicine called BI 456906.

Participants are divided into different groups. All participants in the study either take different doses of BI 1820237 or placebo. Some of the groups take either semaglutide or BI 456906 in addition.

Each participant has an equal chance of being in each group. All participants receive the study medicines as injections under the skin once a week for almost 5 months. Placebo injections look like BI 1820237 injections, but do not contain any medicine. Semaglutide is medicine that is already used for overweight or obesity. BI 456906 is another medicine that is being developed for the treatment of overweight and obesity. Participants are in the study for about 7 months. During this time, they visit the study site regularly. For some of the visits, the participants remain at the study site for 1 or 2 nights. At the study visits, the doctors check the health of the participants and note any health problems that could have been caused by BI 1820237, semaglutide, or BI 456906.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with obesity/overweight (otherwise healthy) according to the assessment of the Investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 27.0 to 40.0 kg/m2 (inclusive). Overweight/obesity should be due to excess adipose tissue, as judged by the Investigator
* Body weight greater than or equal to 75 kg
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Further inclusion criteria apply.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the Investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the Investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the Investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy, bariatric surgery or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of treatment-emergent adverse events | Up to 180 days
  assessed as drug-related by the investigator

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 1820237 in plasma over the time interval from 0 to 168 hours after administration of BI 1820237 or placebo (AUC0-168) | Up to 141 days
Maximum measured concentration of BI 1820237 in plasma (Cmax) | Up to 141 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com